CLINICAL TRIAL: NCT06289283
Title: Profiling Urinary Microbiota In Male Patients With Bladder Cancer
Brief Title: Microbiota in Urine and Urothelium Can be a Factor for Induction of Urinary Bladder Cancer. The Study Will Examine Urine and Bladder Cancer Tissues From Male Patients and Urine of Controls Using Whole Genomic Sequencing Techniques and 16S rRNA. The Aim is to Elucidate Role of Microbiota in Bladder
Acronym: Cancer bladder
Status: Active, not recruiting | Type: Observational
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Mohamed Wishahi, Professor Doctor, Theodor Bilharz Research Institute
Other Study IDs: Theodor Bilharz Research Ins.
Record Dates: First submitted 2024-02-25; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Urinary Bladder Neoplasms; Microtia
MeSH Terms: conditions — Urinary Bladder Neoplasms; Congenital Microtia | interventions — Disinfectants; Preservation, Biological

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine samples and tissue samples of bladder.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bladder carcinoma of non muscle invasive bladder cancer and muscle invasive bladder cancer.: Group I: Non-muscle invasive bladder cancer,16 patients, 16 for bladder tissue, and 16 for urine samples. Total 32 samples. (The study will explore the microbiota in urine and in tissue samples, so every patient with bladder cancer will give (2 samples). The control group will give urine sample ( one samble). Recent research showed that microbiota is detecred in the urothelium of normal undividuals and patients with bladder cancer, this microbiota would differ from urine( liquid) microbiota.(References: ) Group II: Muscle invasive bladder cancer, 11 patients. 22 samples 11 for bladder tissue and 11 for urine samples obtained from the same patients. Group III: 11 Normal adults: urine samples from serves as control group of the study.
  Total number of participant is 38 individual
  Interventions: Other: Urine samples and tissue samples: Samples will be collected in clean leak-proof containers without disinfectant or detergent residue and with tight-fitting leak-proof lids and preserved in a refrigera

INTERVENTIONS:
Other: Urine samples and tissue samples: Samples will be collected in clean leak-proof containers without disinfectant or detergent residue and with tight-fitting leak-proof lids and preserved in a refrigera — Samples for microbiome analysis:
  Samples will be collected in clean leak-proof containers without disinfectant or detergent residue and with tight-fitting leak-proof lids and preserved in a refrigerator until be analyzed at the microbiology laboratory of TBRI.
  Urine samples (50 ml) for microbiome analysis will be collected during cystoscopy examination. Samples will be stored at -80 °C until processing.
  Tissue and urine samples from patients with bladder cancer: Under standard procedure of diagnostic cystoscopy urine sample will be collected under complete aseptic conditions, patients who has bladder tumor will undergo transurethral resection of bladder tumor, a tissue sample 0.5x0.5 cm will be investigated for microbiome analysis. Samples will be stored at -80 °C until processing. Histopathological diagnosis with Hematoxylin and eosin stain will be done by an expert pathologist for tumor grade and stage according to WHO 22, and EAU guidelines 2023. This procedure will be applied for

SUMMARY:
Microbes inhabiting the urinary tract that are playing an important role in maintenance of health and the development of diseases and bladder cancer. There is correlation between initiation of bladder cancer and microbes. Urine and bladder tissues from healthy individuals and patients with bladder cancer were analyzed using 16S rRNA sequencing, results show abundant phylum. Next-generation sequencing technologies will be applied with whole genomic and 16S ribosomal RNA gene sequencing for microbiota profiling in urine and bladder tissue of male healthy individuals and patients with bladder cancer. Results will lead to prevention, diagnosis and new treatment strategies for bladder cancer.

DETAILED DESCRIPTION:
-Rationaly and objectives:

A- Bladder Cancer:

Rationale Bladder cancer is estimated to be the ninth most frequent malignant disease, with 160,000 or more deaths per year estimated globally.

There is an increasingly awareness of the important role of microbes that are inhabiting in the urinary tract that are playing an important role in maintenance of health and the development of diseases and bladder cancer [1].

There is a well-established correlation between initiation of bladder cancer and specific microbial agents [2,3,4,5,].

Damage of the host DNA could be directly initiated via genotoxins produced by specific E. coli strains or via an indirect route by initiating oxidative species. Microbiome and its products have an anticancer effect [6].

Traditionally, urine and bladder urothelium have been considered sterile in healthy individuals. This concept was based on standard microbiological urine cultures. Recently, there is cumulating proofs and evidence that the urinary tract also harbors distinct commensal microorganisms. The urinary microbiome has been reported in healthy individuals [ 7].

The urinary microbiome in bladder cancer has been infrequently investigated, it had been reported that Streptococcus sp was enriched in the bladder of some patients with bladder cancer [8].

Bučević Popović V et al [1] reported that:" Bacterial communities present in urine specimens from male patients with bladder cancer, and from healthy individuals were analyzed using 16S sequencing. The results show that the most abundant phylum in both groups was Firmicutes, followed by Actinobacteria, Bacteroidetes and Proteobacteria. Significantly enriched in the bladder cancer was the genus Fusobacterium, which is a possible protumorigenic pathogen. In bladder cancer tissues, Fusobacterium nucleatum sequences detected by PCR the genera Veillonella, Streptococcus and Corynebacterium were more abundant in healthy urines. Campylobacter hominis was enriched in urine samples of patients with bladder cancer, Campylobacter species are potentially pathogenic as they produce toxins, invades epithelial cells, and can avoid host immune responses".

Microbiota may provide tumor-suppressive effects to the human host [6]. Next-generation sequencing (NGS) technologies has enabled the profiling of microbial communities in specific habitats. 16S ribosomal RNA (rRNA) gene sequencing is used for microbiota profiling with NGS technologies. Choosing which 16S rRNA hypervariable region to sequence is critical in microbiota profiling studies is important. All nine 16S rRNA hypervariable regions are taxonomically informative, but due to variability in profiling performance for specifically, choosing the ideal 16S rRNA hypervariable region will depend on the bacterial composition of the habitat under study. Microbial communities colonizing the urinary tract (the urobiome) are identified in V4,V5. Recent studies have shown that urobiome dysbiosis is linked to several urological conditions [ 9,10,11], and bladder cancer [12].

Objectives: Therefore, it is crucial to characterize the urobiome in health and bladder cancer, and may lead to new prevention, diagnosis and treatment strategies for bladder cancer.

Objectives The aim of this research study is to characterize the urinary microbiota of adult male patients with bladder cancer and to be correlated with microbiota in healthy adult males controls.

2-Methodology 2-1 Study type: Prospective case control study 2-2 Inclusion, exclusion criteria, recruitment process. [ included patients in the study will be asked to offer an informed consent, Dr Loay Mostafa and Dr. Mohamed Sahab from the Urology Department - TBRI will be responsible for this item].

Inclusion Criteria:

* Adult men above 18 years,
* Diagnosed of carcinoma of the bladder with imaging ultrasonography and/ or computerized tomography, and urine cytology.
* Confirmed bladder cancer either during diagnostic cystoscopy, previous pathology, or pathological examination of the biopsy specimens.

Exclusion criteria:

* Previous radiotherapy to the bladder or to adjacent organ.
* Previous intravesical instillation immunotherapy with bacillus Calmette-Guérin (BCG), or intravesical instillation of chemotherapeutics.
* Previous neoadjuvant chemotherapy. Recruitment process Patients fulfilling the exclusion and inclusion criteria. 2-3 Sample size Thirty eight Egyptian men, age ≥ 18, will be recruited at the Department of Urology, TBRI according to sample size calculation using online software (Sample Size Calculator). Ten urine samples will be collected from normal individuals.

https://www.calculator.net/sample-size-calculator.html Sample size will be 16 for non-muscle invasive bladder cancer (NMIBC). This means 16 or more measurements/surveys are needed to have a confidence level of 95%. Sample size will be 11 for muscle invasive bladder cancer (MIBC). This means 40 or more measurements/surveys are needed to have a confidence level of 95%. Sample size will be 11 for control group. This means 10 or more measurements/surveys are needed to have a confidence level of 95% A. 38 men will be recruited at the Department of Urology, TBRI. According to sample size calculation using online software (Sample Size Calculator). Eleven urine samples will be collected from Sample size will be 16 for non-muscle invasive bladder cancer (NMIBC). This means 16 or more measurements/surveys are needed to have a confidence level of 95% that the real value is within ±17.53% of the measured/surveyed value.

Sample size will be 11 for muscle invasive bladder cancer (MIBC). This means 11 or more measurements/surveys are needed to have a confidence level of 95% that the real value is within ±30.36% of the measured/surveyed value.

Sample size will be 11 for control group. This means 11 or more measurements/surveys are needed to have a confidence level of 95% that the real value is within ±30.36% of the measured/surveyed value.

normal individuals. This sample represents the research on microbiome in bladder cancer.

https://www.calculator.net/sample-size-calculator.html 2-4 Sample collection

Bladder cancer:

The total number of studied samples: The study will explore the microbiota in urine and in tissue samples, so every patient with bladder cancer will give (2 samples). The control group will give urine sample ( one samble). Recent research showed that microbiota is detecred in the urothelium of normal undividuals and patients with bladder cancer, this microbiota would differ from urine( liquid) microbiota.

References:

1. Mansour B, Monyók Á, Makra N, Gajdács M, Vadnay I, Ligeti B, Juhász J, Szabó D, Ostorházi E. Bladder cancer-related microbiota: examining differences in urine and tissue samples. Sci Rep. 2020 Jul 6;10(1):11042. doi: 10.1038/s41598-020-67443-2.
2. Parra-Grande M, Oré-Arce M, Martínez-Priego L, D'Auria G, Rosselló-Mora R, Lillo M, Sempere A, Lumbreras B, Sánchez-Hellín V. Profiling the Bladder Microbiota in Patients With Bladder Cancer. Front Microbiol. 2022 Feb 7;12:718776. doi: 10.3389/fmicb.2021.718776.

   Group I: Non-muscle invasive bladder cancer,16 patients, 16 for bladder tissue, and 16 for urine samples. Total 32 samples. (The study will explore the microbiota in urine and in tissue samples, so every patient with bladder cancer will give (2 samples). The control group will give urine sample ( one samble). Recent research showed that microbiota is detecred in the urothelium of normal undividuals and patients with bladder cancer, this microbiota would differ from urine( liquid) microbiota.(References: ) Group II: Muscle invasive bladder cancer, 11 patients. 22 samples 11 for bladder tissue and 11 for urine samples obtained from the same patients. Group III: 11 Normal adults: urine samples from serves as control group of the study.

   Total number of participant is 38 individual.

   Samples for microbiome analysis:

   Samples will be collected in clean leak-proof containers without disinfectant or detergent residue and with tight-fitting leak-proof lids and preserved in a refrigerator until be analyzed at the microbiology laboratory of TBRI.

   Urine samples (50 ml) for microbiome analysis will be collected during cystoscopy examination. Samples will be stored at -80 °C until processing.

   Tissue and urine samples from patients with bladder cancer: Under standard procedure of diagnostic cystoscopy urine sample will be collected under complete aseptic conditions, patients who has bladder tumor will undergo transurethral resection of bladder tumor, a tissue sample 0.5x0.5 cm will be investigated for microbiome analysis. Samples will be stored at -80 °C until processing. Histopathological diagnosis with Hematoxylin and eosin stain will be done by an expert pathologist for tumor grade and stage according to WHO 22, and EAU guidelines 2023. This procedure will be applied for both non-muscle invasive and muscle invasive urothelial carcinoma. Patients who will undergo radical cystectomy for bladder cancer will be included in the sample size.

   Samples for pathological studies:

   Tissue samples will be fixed with formalin and examined with hematoxylin and eosin stain.

   Clinical Information The urologists will provide adequate tissue samples which is a small part of the whole resected tumor or a part of cystectomy specimens. for pathological evaluation with giving useful clinical information to the pathologist to decide the best approach in handling and processing the surgical specimens and draw up an accurate pathology report.

   The urologist will specify:
   * Demographic data and clinical history of the patient, history of urinary tract infection and if it was recurrent or sporadic, bladder cytology if present, whether it is the first presentation of the tumor and if not, details of previous management.
   * The cystoscopic appearance of bladder mucosa and indicate number, size, location of the tumor/s, the morphological features of the lesion: papillary, solid, or ulcerate.
   * The state of remaining mucosa if further biopsies were performed.

   Theses information is necessary for a correct evaluation of urothelium and search in microbiome. Because the treatments can have an impact on tumor morphology and on normal looking urothelium.

   Bladder Cancer Samples Reporting
   * Pathological assessment The pathologist will diagnose if a bladder cancer is present and the type of bladder cancer, by examining cells from the bladder tissue biopsy. Different histological tumor types of bladder cancer will be reported according to the 2016 WHO classification of urinary bladder tumors (Mazzucchelli et al. 2021), modified in 2022.
   * Microbiological assessment: Microbial identification methods from Urine and tissue

   Sample collection and culture conditions of clinical bacterial isolates:

   Detection of a limited number of microorganisms, mainly aerobic and fast-growing bacteria.

   Identification of bacterial isolates: The isolates will be identified by culturing on blood, MacConkey agar and sabaruds agar then will be identified by performing biochemical tests, oxidase test mannitol, bile esculin, and catalase test. All isolates will be identified to species level by using Vitek 2 compact system.

   2-5 Biochemestry and molecular biology assessment: 16S Metagenomic Sequencing analysis Whole genomic sequencing (WGS) will be applied to all cases, methodology and quality control are according to the genomic and metagenomic center in the children cancer hospital 57357 who are going to perform the WGS and 16S sequencing on urine and tissue samples.

1- DNA isolation from urine and tissue. Urine specimens (50ml) will be thawed and centrifuged at 7500g, 4°C for 10minutes. The pellet will be used for DNA extraction using Invitrogen™ PureLink™ Microbiome DNA Purification Kit, performed according to manufacturer's protocol. To avoid environmental contamination, all isolations from urine samples and from the reagent-only extraction control will be carried out within a PCR hood. Isolated DNA samples will be placed at -20 °C until PCR amplifcation. DNA will be quantifed using DeNovix dsDNA High Sensitivity Assay Kit (Illumina 2013) .

2- PCR based KABA KAPA Library Quantification Kits contain all the reagents needed for the accurate, reliable and reproducible qPCR-based quantification of next-generation sequencing (NGS) libraries prepared for sequencing on Illumina platforms. Kits include KAPA SYBR FAST qPCR Master Mix (formulated with different passive reference dyes for different qPCR instruments), a platform- specific library quantification primer premix, and a pre-diluted set of DNA standards.

16S rRNA gene V3-V4 region will be amplifed with fusion primers that incorporate Illumina adapters and indexing barcodes. The PCR step adds Index 1 (i7) and Index 2 (i5), sequencing, and common adapters (P5 and P7) required for cluster generation and sequencing. High Sensitivity DNA electrophoresis with the Bioanalyzer system will be done to improve quality control analysis of NGS library. 3- 16S rRNA gene library preparation and MiSeq sequencing. PCR amplification of 16S rDNA, sequencing and analyses will be performed by NGS Illumina MiSeq targeting V3V4 region of bacteria MiSeq Reagent Kit v3 (600-cycle). 16S rRNA gene amplicon sequencing (16S analysis) is widely used to analyze microbiota with next-generation sequencing technologies. 16S analysis data from the standard V3-V4 primer (V34) sets to optimize the bladder microbiota analysis protocol. 4- Bioinformatics and statistical analyses. The annotated genome is further analyzed using bioinformatic pipelines to gain insights into the pathogen's biology and potential for causing disease. It includes:

- Quality control and improvement of the draft genome by removing errors and filling in gaps.

* Annotation of the final genome, including identifying and describing the functions of genes and other features.
* Comparative genomics, which involves comparing the newly sequenced genome to those of related pathogens to identify differences and similarities.
* Functional analysis: this involves identifying the functions of the annotated genes and understanding the pathways and processes they participate in. This can reveal key virulence factors and help to understand the pathogen's pathogenesis mechanism.
* Phylogenetic analysis: This involves comparing the newly sequenced genome to those of
* related pathogens to determine evolutionary relationships and track the spread of pathogens in different populations.
* Differences in the overall microbial composition between bladder cancer and healthy
* samples will be assessed. NGS is not available in TBRI, the 16S sequencing and bioinformatics will be done paid in Children Hospital 57357 (they are welcomed to perform the sequencing on a"Paid" principle).

  16S ribosomal RNA (rRNA)Sequencing analysis
  1. DNA isolation from urine and tissue. Urine specimens (50ml) will be thawed and centrifuged at 7500g, 4°C for 10minutes. The pellet will be used for DNA extraction using microbiome DNA Purification Kit. To avoid environmental contamination, all isolations from urine samples and from the reagent-only extraction control will be carried out within a PCR hood. Isolated DNA samples will be placed at -20 °C until PCR amplification. DNA will be quantified using an assay Kit (Illumina 2013).
  2. PCR based KABA KAPA Library Quantification Kits contain all the reagents needed for the accurate, reliable and reproducible qPCR-based quantification of next-generation sequencing (NGS) libraries prepared for sequencing on Illumina platforms. A platform-specific library quantification primer premix, and a pre-diluted set of DNA standards.

  16S rRNA hypervariable regionsV1V2 and V3-V4 region will be amplifed with fusion primers that incorporate Illumina adapters and indexing barcodes.

High Sensitivity DNA electrophoresis with the Bioanalyzer system will be done to improve quality control analysis of NGS library.

3- 16S rRNA gene library preparation and MiSeq sequencing. PCR amplification of 16S rRNA, sequencing and analyses will be performed by NGS Illumina targeting V1-V2 and V3-V4 region. 16S rRNA gene amplicon sequencing (16S analysis) will be used to analyze microbiota with next-generation sequencing technologies. 16S analysis data from the standard V1-V2, V3-V4 primer sets to optimize the bladder microbiota analysis protocol.

4- Bioinformatics and statistical analyses. The annotated genome is further analyzed using bioinformatic pipelines to gain insights into the pathogen's biology and potential for causing disease.

References

1. Bučević Popović V, Šitum M, Chow CT, Chan LS, Roje B, Terzić J. The urinary microbiome associated with bladder cancer. Sci Rep. 2018 Aug 14;8(1):12157. doi: 10.1038/s41598-018-29054-w.
2. Wishahi, M., Otto, T. & Golka, K. Re: bladder carcinomas in patients with neurogenic bladder and urinary schistosomiasis-are they the same tumors?. World J Urol 40, 2139-2140 (2022). https://doi.org/10.1007/s00345-022-04076-2
3. Hanan R, Murata M, Ma N, Hammam O, Wishahi M, El Leithy T, Hiraku Y, Oikawa S, Kawanishi S (2012) Nuclear localization of COX-2 in relation to the expression of stemness markers in urinary bladder cancer. Mediat Inflamm 2012:165879 2012;2012:165879. doi: 10.1155/2012/165879.
4. Cancrini F, Michel F, Cussenot O, Alshehhi H, Comperat E, Phé V (2022) Bladder carcinomas in patients with neurogenic bladder and urinary schistosomiasis: are they the same tumors? World J Urol. https://doi.org/10.1007/s00345-022-03941-4
5. Hammam O, Wishahi M, Khalil H, El Ganzouri H, Badawy M, Elkhquly A, Elesaily K (2014) Expression of cytokeratin 7, 20, 14 in urothelial carcinoma and squamous cell carcinoma of the Egyptian urinary bladder cancer. J Egypt Soc Parasitol 44(3):733-740
6. Zitvogel L, Daillère R, Roberti MP, Routy B, Kroemer G. Anticancer effects of the microbiome and its products. Nat. Rev. Microbiol. 2017;15:109-128. doi: 10.1038/nrmicro.2017.44.
7. Whiteside SA, Razvi H, Dave S, Reid G, Burton JP. The microbiome of the urinary tract - a role beyond infection. Nat. Rev. Urol. 2015;12:81-90. doi: 10.1038/nrurol.2014.361.
8. Xu W, et al. Mini-review: perspective of the microbiome in the pathogenesis of urothelial carcinoma. Am. J. Clin. Exp. Urol. 2014;2:57-61.
9. Brubaker, L., Gourdine, J.-P. F., Siddiqui, N. Y., Holland, A., Halverson, T., Limeria, R., et al. (2021a). Forming Consensus To Advance Urobiome Research. mSystems 6, e0137120. doi: 10.1128/mSystems.01371-20
10. Brubaker, L., Putonti, C., Dong, Q., and Wolfe, A. J. (2021b). The Human Urobiome. Mamm. Genome 32, 232-238. doi: 10.1007/s00335-021-09862-8
11. -Carrasco, V., Soriano-Lerma, A., Soriano, M., J., and Garcia-Salcedo, J. A. (2021). Urinary Microbiome: Yin and Yang of the Urinary Tract. Front. Cell. Infect. Microbiol. 11. doi: 10.3389/fcimb.2021.617002
12. 43. Wu N, et al. Dysbiosis signature of fecal microbiota in colorectal cancer patients. Microb. Ecol. 2013;66:462-470. doi: 10.1007/s00248-013-0245-9.

ELIGIBILITY:
Inclusion Criteria:

* Adult men above 18 years,
* Diagnosed of carcinoma of the bladder with imaging ultrasonography and/ or computerized tomography, and urine cytology.
* Confirmed bladder cancer either during diagnostic cystoscopy, previous pathology, or pathological examination of the biopsy specimens.

Exclusion criteria:

* Previous radiotherapy to the bladder or to adjacent organ.
* Previous intravesical instillation immunotherapy with bacillus Calmette-Guérin (BCG), or intravesical instillation of chemotherapeutics.
* Previous neoadjuvant chemotherapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group I: Non-muscle invasive bladder cancer,16 patients, 16 for bladder tissue, and 16 for urine samples. Total 32 samples. (The study will explore the microbiota in urine and in tissue samples, so every patient with bladder cancer will give (2 samples). The control group will give urine sample ( one samble). ) Group II: Muscle invasive bladder cancer, 11 patients. 22 samples 11 for bladder tissue and 11 for urine samples obtained from the same patients. Group III: 11 Normal adults: urine samples from serves as control group of the study.
  Total number of participant is 38 individual.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To characterize the microbiota in health and bladder cancer, and may lead to new prevention, diagnosis and treatment strategies for bladder cancer | Sample sollection 12 months, next generation sequencing ind bioinformatics 6 months, interpretation of data 6 months.
  Biochemestry and molecular biology assessment: 16S Metagenomic Sequencing analysis Whole genomic sequencing (WGS) will be applied to all cases, methodology and quality control are according to the genomic and metagenomic center in the children cancer hospital 57357 who are going to perform the WGS and 16S sequencing on urine and tissue samples. 1- DNA isolation from urine and tissue. Urine specimens (50ml) will be thawed and centrifuged at 7500g, 4°C for 10minutes. The pellet will be used for DNA extraction using Invitrogen™ PureLink™ Microbiome DNA Purification Kit, performed according to manufacturer's protocol. To avoid environmental contamination, all isolations from urine samples and from the reagent-only extraction control will be carried out within a PCR hood. Isolated DNA samples will be placed at -20 °C until PCR amplifcation. DNA will be quantifed using DeNovix dsDNA High Sensitivity Assay Kit (Illumina 2013) . 2- PCR based KABA KAPA Library Quantification Kits contain all

CONTACTS AND LOCATIONS:
Locations (1):
- Theodor Bilharz Research Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Decision will be after the study will be finished and data analysis.

REFERENCES:
- [Background] Whiteside SA, Razvi H, Dave S, Reid G, Burton JP. The microbiome of the urinary tract--a role beyond infection. Nat Rev Urol. 2015 Feb;12(2):81-90. doi: 10.1038/nrurol.2014.361. Epub 2015 Jan 20. PMID 25600098